CLINICAL TRIAL: NCT02497105
Title: Ketogenic Diet Program for Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: University of Hawaii (Other)
Responsible Party: Principal Investigator, Ryan Lee, MD, Director - Neurodevelopmental Clinic, Research, Shriners Hospitals for Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HON1402
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Epilepsy
Keywords: Epilepsy; Intractable Seizures; Ketogenic Diet; Biochemical Profiles
MeSH Terms: conditions — Epilepsy | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epilepsy/Ketogenic Diet (Experimental): Children (0-18 years of age) diagnosed with epilepsy will receive the ketogenic diet intervention.
  Interventions: Other: Ketogenic Diet
- Epilepsy/Non-Ketogenic Diet (No Intervention): Children (0-18 years of age) diagnosed with epilepsy will not receive the ketogenic diet intervention.

INTERVENTIONS:
Other: Ketogenic Diet — Dietary
  Arms: Epilepsy/Ketogenic Diet

SUMMARY:
This study will assess the effectiveness of the ketogenic diet (high-fat, low-carbohydrate, and moderate protein) in treating epilepsy. Two study groups will be comprised of children with epilepsy (0-18 years of age) and whether or not they receive the ketogenic diet - epilepsy/ketogenic diet and epilepsy/non-ketogenic diet.

DETAILED DESCRIPTION:
According to an evidence-based guideline on the diagnosis and management of epilepsy from the National Institute for Clinical Excellence (2012), the ketogenic diet may be considered as an adjunctive treatment in children with drug-resistant epilepsy. Vast anecdotal and Class 1 studies have confirmed that the ketogenic diet helps most children with intractable seizures and cures many. Dietary therapies for epilepsy (e.g., classic ketogenic diet) have been shown to be highly effective. For example, Lee (P.R.) and Kossoff reported that approximately 50% of children with drug-resistant epilepsy had a greater than 50% reduction in seizures within days to months of treatment. In addition, use of the ketogenic diet as a treatment for epilepsy has been shown to reduce the escalating costs associated managing poorly controlled seizures (e.g., decrease in outpatient and emergency visits, inpatient hospitalization, neuroimaging, electro-encephalography, lab testing, and medication use).

If a child's seizures continue after two to three seizure medications have been tried, the ketogenic diet should be considered. However, many parents still medicate their children well beyond these guidelines and tolerate seizure frequency because they have no other alternatives. Given the physical and emotional toll that recurring seizures exact upon these children/families, the potential for improvement with the ketogenic diet is substantial. However, the ketogenic diet remains unavailable to most children.

Approximately 1% of Hawaii's children are projected to have epilepsy, but there is no established, ketogenic diet program for them to receive this dietary intervention, which can incorporate culturally distinct foods to improve palatability and compliance. Although the ketogenic diet has shown promise for broadening the scope of therapeutic options for children with epilepsy, it requires further study in an ethnically diverse population. At Shriners Hospitals for Children-Honolulu, the investigators have initiated a ketogenic and related dietary (e.g., modified Atkins diet) intervention program for children with epilepsy and started to assess its efficacy in treating epilepsy/seizures. This program also includes educational seminars and services to patients residing on the other Hawaii islands through outreach trips. The investigators have begun to enroll children with epilepsy into two groups based on whether or not they receive the ketogenic diet - epilepsy/ketogenic diet and epilepsy/non-ketogenic diet; total estimate of 15-30 participants over three years. Based upon initial findings, the investigators will implement a comprehensive, multidisciplinary ketogenic diet program that will potentially reach hundreds of children throughout Hawaii, the Pacific Basin, and elsewhere.

Specific Aims:

Aim 1. To assess the therapeutic efficacy of the ketogenic diet on epilepsy/seizures.

Hypothesis: Participants who have epilepsy/on the ketogenic diet will have significantly decreased number and severity of seizures than those that are not on the ketogenic diet, between baseline to three and six months after the dietary intervention is initiated.

Aim 2. In anticipation of lessened epilepsy/seizures, to determine the (a) change in number and dose of seizure medications used, (b) change in number of lab tests ordered for epilepsy management, (c) change in number of emergency room and hospital visits for seizures (or other neurodevelopmental problems), (d) change in number of neurologic procedures for epilepsy management (e.g. EEG, MRI, CT), and (e) participant/family satisfaction with the ketogenic diet.

Hypothesis: The number and/or dosage of medications, lab tests ordered, emergency room or hospital visits, and neurologic procedures for epilepsy management will decrease, and participant/family satisfaction will be high for participants who have epilepsy/on the ketogenic diet than those that are not on the ketogenic diet, between baseline to three and six months after the dietary intervention is initiated.

Aim 3. To compare differences and/or changes in (a) serum and urine ketone levels and (b) biochemical profiles as defined from blood and stool (gut or fecal microbiome) specimen samples.

Hypothesis: Participants who have epilepsy/on the ketogenic diet will have significantly higher serum/urine ketone levels and notably different biochemical profiles than those that are not on the ketogenic diet, between baseline to three and six months after the dietary intervention is initiated.

Children helped by the ketogenic diet are more likely to reach their highest level of functioning and become contributing adults. By providing the ketogenic diet as an intervention therapy for epilepsy in a safe and data-driven manner, the community-at-large will benefit and medical knowledge concerning dietary treatment for neurodevelopmental disorders will be advanced.

ELIGIBILITY:
Inclusion Criteria:

* Ages 0-18 years.
* Primary diagnosis of epilepsy.
* Parent/legal guardian and child able to read or understand English, and able/willing to provide informed consent/assent.
* Females of childbearing potential must have a negative pregnancy test result and agree to use a medically acceptable method of contraception throughout the entire study period and for 30 days after the last dose of study drug - childbearing potential is defined a girls who are > Tanner stage 2 and urine pregnancy tests are acceptable.

Exclusion Criteria:

* Known cardiac disorder including arrhythmias or hypertension.
* Carnitine deficiency (primary).
* Carnitine palmitoyltransferase (CPT) I or II deficiency.
* Carnitine translocase deficiency.
* Beta-oxidation defects - medium-chain acyl dehydrogenase deficiency (MCAD), long-chain acyl dehydrogenase deficiency (LCAD), short-chain acyld dehydrogenase deficiency (SCAD), long-chain 3-hydroxyacyl-coenzyme A (CoA) deficiency, and medium-chain 3-hydroxyacyl-CoA deficiency.
* Pyruvate carboxylase deficiency.
* Porphyria.
* Inability to maintain adequate nutrition.
* Patient or caregiver non-compliance.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the core symptoms of epilepsy (seizure frequency/severity) | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess the number of epileptic seizures through review/analysis of responses to the seizure log (self-report)

SECONDARY OUTCOMES:
Change from baseline in the number of medications used for epilepsy management | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess changes through the review/analysis of self-report and medical record data
Change from baseline in the dosage of medications used for epilepsy management | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess changes through the review/analysis of self-report and medical record data
Change from baseline in the number of lab tests ordered for epilepsy management | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess changes through the review/analysis of self-report and medical record data
Change from baseline in the number of emergency room or hospital visits for epilepsy management | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess changes through the review/analysis of self-report and medical record data
Change from baseline in subject/family satisfaction with the ketogenic diet | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess changes through the review/analysis of self-report and medical record data
Change from baseline in ketone levels due to the ketogenic diet | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess ketone level differences and changes through the analysis of serum and urine
Change from baseline in biochemical profiles due to the ketogenic diet | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess biochemical profile differences and changes through the analysis of blood and stool (gut microbiome) specimen samples

CONTACTS AND LOCATIONS:
Overall Officials: Ryan W Lee, MD, Principal Investigator — Shriners Hospitals for Children, Honolulu
Locations (1):
- Shriners Hospitals for Children - Honolulu, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] http://www.aetna.com/cpb/medical/data/200_299/0226.html Clinical Policy Bulletin: Hospitalization for the Initiation of Ketogenic Diet for the Treatment of Intractable Seizures. Accessed November 14, 2013.
- [Background] Cervenka MC, Kossoff EH. Dietary treatment of intractable epilepsy. Continuum (Minneap Minn). 2013 Jun;19(3 Epilepsy):756-66. doi: 10.1212/01.CON.0000431396.23852.56. PMID 23739109
- [Background] National Clinical Guideline Centre (UK). The Epilepsies: The Diagnosis and Management of the Epilepsies in Adults and Children in Primary and Secondary Care: Pharmacological Update of Clinical Guideline 20. London: Royal College of Physicians (UK); 2012 Jan. Available from http://www.ncbi.nlm.nih.gov/books/NBK247130/ PMID 25340221
- [Background] http://www.charliefoundation.org/offering-hope.html Accessed November 14, 2013
- [Background] Lee PR, Kossoff EH. Dietary treatments for epilepsy: management guidelines for the general practitioner. Epilepsy Behav. 2011 Jun;21(2):115-21. doi: 10.1016/j.yebeh.2011.03.008. Epub 2011 Apr 21. PMID 21514240
- [Background] Williams E, Abrahams J, Maguire A, Harris G. A parent's perspective on dietary treatments for epilepsy. Epilepsy Res. 2012 Jul;100(3):338-43. doi: 10.1016/j.eplepsyres.2011.09.024. Epub 2012 May 8. PMID 22575229
- [Background] Kossoff EH, Caraballo RH, du Toit T, Kim HD, MacKay MT, Nathan JK, Philip SG. Dietary therapies: a worldwide phenomenon. Epilepsy Res. 2012 Jul;100(3):205-9. doi: 10.1016/j.eplepsyres.2011.05.024. PMID 21856128
- [Background] Gilbert DL, Pyzik PL, Vining EP, Freeman JM. Medication cost reduction in children on the ketogenic diet: data from a prospective study. J Child Neurol. 1999 Jul;14(7):469-71. doi: 10.1177/088307389901400712. PMID 10573471
- [Background] Mandel A, Ballew M, Pina-Garza JE, Stalmasek V, Clemens LH. Medical costs are reduced when children with intractable epilepsy are successfully treated with the ketogenic diet. J Am Diet Assoc. 2002 Mar;102(3):396-8. doi: 10.1016/s0002-8223(02)90091-x. PMID 11902372
- [Background] Vining EP, Freeman JM, Ballaban-Gil K, Camfield CS, Camfield PR, Holmes GL, Shinnar S, Shuman R, Trevathan E, Wheless JW. A multicenter study of the efficacy of the ketogenic diet. Arch Neurol. 1998 Nov;55(11):1433-7. doi: 10.1001/archneur.55.11.1433. PMID 9823827
- [Background] Freeman JM, Vining EP, Pillas DJ, Pyzik PL, Casey JC, Kelly LM. The efficacy of the ketogenic diet-1998: a prospective evaluation of intervention in 150 children. Pediatrics. 1998 Dec;102(6):1358-63. doi: 10.1542/peds.102.6.1358. PMID 9832569
- [Background] Neal EG, Chaffe H, Schwartz RH, Lawson MS, Edwards N, Fitzsimmons G, Whitney A, Cross JH. The ketogenic diet for the treatment of childhood epilepsy: a randomised controlled trial. Lancet Neurol. 2008 Jun;7(6):500-6. doi: 10.1016/S1474-4422(08)70092-9. Epub 2008 May 2. PMID 18456557
- [Background] Henderson CB, Filloux FM, Alder SC, Lyon JL, Caplin DA. Efficacy of the ketogenic diet as a treatment option for epilepsy: meta-analysis. J Child Neurol. 2006 Mar;21(3):193-8. doi: 10.2310/7010.2006.00044. PMID 16901419
- [Background] Beghi E, Frigeni B, Beghi M, De Compadri P, Garattini L. A review of the costs of managing childhood epilepsy. Pharmacoeconomics. 2005;23(1):27-45. doi: 10.2165/00019053-200523010-00003. PMID 15693726
- [Background] de Kinderen RJ, Lambrechts DA, Postulart D, Kessels AG, Hendriksen JG, Aldenkamp AP, Evers SM, Majoie MH. Research into the (Cost-) effectiveness of the ketogenic diet among children and adolescents with intractable epilepsy: design of a randomized controlled trial. BMC Neurol. 2011 Jan 25;11:10. doi: 10.1186/1471-2377-11-10. PMID 21262002
- [Background] Herbert MR, Buckley JA. Autism and dietary therapy: case report and review of the literature. J Child Neurol. 2013 Aug;28(8):975-82. doi: 10.1177/0883073813488668. Epub 2013 May 10. PMID 23666039
- [Background] De Angelis M, Piccolo M, Vannini L, Siragusa S, De Giacomo A, Serrazzanetti DI, Cristofori F, Guerzoni ME, Gobbetti M, Francavilla R. Fecal microbiota and metabolome of children with autism and pervasive developmental disorder not otherwise specified. PLoS One. 2013 Oct 9;8(10):e76993. doi: 10.1371/journal.pone.0076993. eCollection 2013. PMID 24130822
- [Background] Kossoff EH, Zupec-Kania BA, Amark PE, Ballaban-Gil KR, Christina Bergqvist AG, Blackford R, Buchhalter JR, Caraballo RH, Helen Cross J, Dahlin MG, Donner EJ, Klepper J, Jehle RS, Kim HD, Christiana Liu YM, Nation J, Nordli DR Jr, Pfeifer HH, Rho JM, Stafstrom CE, Thiele EA, Turner Z, Wirrell EC, Wheless JW, Veggiotti P, Vining EP; Charlie Foundation, Practice Committee of the Child Neurology Society; Practice Committee of the Child Neurology Society; International Ketogenic Diet Study Group. Optimal clinical management of children receiving the ketogenic diet: recommendations of the International Ketogenic Diet Study Group. Epilepsia. 2009 Feb;50(2):304-17. doi: 10.1111/j.1528-1167.2008.01765.x. Epub 2008 Sep 23. PMID 18823325
- [Background] Milani C, Hevia A, Foroni E, Duranti S, Turroni F, Lugli GA, Sanchez B, Martin R, Gueimonde M, van Sinderen D, Margolles A, Ventura M. Assessing the fecal microbiota: an optimized ion torrent 16S rRNA gene-based analysis protocol. PLoS One. 2013 Jul 15;8(7):e68739. doi: 10.1371/journal.pone.0068739. Print 2013. PMID 23869230